CLINICAL TRIAL: NCT01753804
Title: A Prospective Natural History Study of Progression of Physical Impairment, Activity Limitation and Quality of Life in Duchenne Muscular Dystrophy.
Brief Title: A Prospective Natural History Study of Progression of Subjects With Duchenne Muscular Dystrophy.
Status: Terminated | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-DMD-01
Record Dates: First submitted 2012-12-13; First posted 2012-12-20 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Myopathy; Natural History; Muscular dystrophy; Biomarkers; Muscle testing
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Diseases; Muscular Dystrophies | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling at 4 time points (first visit then once a year). Urinalysis sampling at 4 time points (first visit then once a year).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study participants: All participants will follow the same protocol, including muscle strength and function testing, and blood and urine collection, for a maximum of 7 visits over 3 years.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — There is no medication or device tested in this study. This is an obversational study on the progression of the disease.

SUMMARY:
To characterize the natural history and progression of Duchenne Muscular Dystrophy (DMD) to help inform the design of future studies, to capture biomarkers of safety and disease progression and to provide comparative data for the development of rare exons for which formal controlled trials are not feasible.

DETAILED DESCRIPTION:
This is a prospective study. All DMD patients that fulfil the inclusion/exclusion criteria are eligible although the study is weighted towards ambulant subjects aged 3 years or older. There will be 7 study visits and subjects will be in the study for a maximum of 3 years. Visits will occur every 6 months (+/- 1 month).

Up to 250 DMD subjects planned in the following categories :

* 75 % ambulant subjects aged between 3 and 18 years at study entry
* 25% non-ambulant subjects with a maximum age of 18 years at study entry

Subjects will be asked to perform muscle testing assessment with a clinical evaluator, such as walking for 6 minutes, climb stairs, breathe in a tube, see how they can move their arms and legs. They will be asked questions about how they feel overall and perform daily activities. These measurements will be assessed every 6 months.

Urine and blood samples will be collected once a year to measure biomarkers that will allow to have a better overview of DMD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD resulting from a mutation in the DMD gene confirmed by a state of the art DNA diagnostic technique covering all DMD gene exons.
* Age 3 - 18 years
* Willing and able to comply with protocol requirements
* Life expectancy of at least 3 years
* Able to give informed assent and/or consent in writing signed by the subject and/or parent(s)/legal guardian (according to local regulations)

Exclusion Criteria:

* Current participation in a clinical study with an Investigational Medicinal Product (IMP)
* Participation within the previous 1 month in a clinical study with an IMP

Ages: 3 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects diagnosed with DMD resulting from a mutation in the DMD gene which is confirmed by a state of the art DNA diagnostic technique covering all DMD gene exons
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
6 minute walk distance | Change from visit 1 walking distance
  Participants are asked to walk at their own preferred speed on a fixed distance for 6 minutes. Subjects are warned of the time and that they may stop earlier if they feel unable to continue. Total distance walked within 6 minutes (or until stopping) is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Goemans, MD, Principal Investigator — UZ Leuven, Belgium
Locations (16):
- United States (3):
  - UC Davis Health System, Sacramento, California
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
- Hospital de Pediatria Prof Dr Juan P Garrahan, Buenos Aires, Argentina
- Belgium (2):
  - Universitair Ziekenhuis, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
- Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, Brazil
- CHU Hopital des enfants, Toulouse, France
- Germany (2):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- Italy (2):
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Policlinico Univsersitario Agostino Gemelli, Rome
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - UMC St. Radboud, Nijmegen
- Drottning Silvias Barn- ochungdomssjukhus, Gothenburg, Sweden
- Hacettepe University Medical Faculty, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: BioMarin website — http://www.biomarin.com